CLINICAL TRIAL: NCT03824275
Title: 18F-DCFPyL Positron Emission Tomography (PET)/Computed Tomography (CT) in Men With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Matthew Dallos, Associate Clinical Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAS1862
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F- DCFPyL PET/CT (Experimental): Upon enrollment, subjects will undergo standard of care imaging (defined as a CT or MRI of the chest, abdomen, and pelvis, and 99mTc bone scans) if not obtained within 45 days of enrollment. Subjects will have standard of care laboratory evaluations including complete blood count (CBC), serum chemistries, hepatic panel, lactate dehydrogenase (LDH), and PSA. Liquid biopsies for circulating tumor DNA (ctDNA) and exosome analysis will occur at the same time. Subjects will then undergo 18F- DCFPyL PET/CT.
  Interventions: Drug: 18F- DCFPyL PET/CT

INTERVENTIONS:
Drug: 18F- DCFPyL PET/CT — A CT scan using a radioactive marker to better image tumors
  Other Names: CT scan

SUMMARY:
PyL, also known as [18F]DCFPyL, is a second-generation fluorinated prostate-specific membrane antigen (PSMA) targeted PET imaging agent. In preliminary studies it demonstrates a higher detection of metastatic prostate lesions compared to standard imaging. Its ability to image metastatic prostate cancer sites was comparable to 68Ga-PSMA with high tumor-to-background ratios.Additionally, [18F] PyL demonstrated higher mean tumor-to-background ratios when using kidney, spleen, or parotid as reference organs. However, the role of [18F] PyL in tumor response to therapy has not been evaluated, specifically the potential to serve as a predictive biomarker of response. Given the high cost of current therapeutic agents in mCRPC, there is a need for an early response biomarker to stratify which patients will benefit from therapy and which will not. This will also allow for earlier change in management of patients who will not response to these therapies, potentially improving patient outcomes.

DETAILED DESCRIPTION:
The investigators will conduct a prospective phase II/III study of 300 men diagnosed with prostate cancer with a rising prostate-specific antigen (PSA). Upon enrollment, subjects will undergo standard of care imaging (defined as a CT or MRI of the chest, abdomen, and pelvis, and 99mTc bone scans) if not obtained within 45 days of enrollment. Subjects will have standard of care laboratory evaluations and undergo 18F- DCFPyL PET/CT.

[18F]DCFPyL will be used for study imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of prostate cancer
2. PSA ≥ 0.2ng/ml
3. Age ≥ 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (karnofsky ≥ 60%)
5. Ability to understand and willingness to sign a written informed consent document
6. Wiling to comply with clinical trial instructions and requirements
7. Willing to cover the cost of PyL PET/CT imaging if funds are not available

Exclusion Criteria:

1. History of another active malignancy within 3 years, other than basal cell and squamous cell carcinoma of the skin
2. Presence of prostate brachytherapy implants unless approved by the PI
3. Administration of another radioisotope within five physical half-lives of trial enrollment
4. Radiation or chemotherapy within 2 weeks prior to trial enrollment
5. Serum creatinine > 3 times the upper limit of normal
6. Serum total bilirubin > 3 times the upper limit of normal
7. Aspartate transaminase (AST) or alanine aminotransferase (ALT) >5 times the upper limit of normal
8. Inadequate venous access

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To determine the positive predictive value of 18F-DCFPyL PET/CT on a per-patient basis | 3.5 years
  To determine the positive predictive value of 18F-DCFPyL PET/CT on a per-patient basis

SECONDARY OUTCOMES:
To determine the positive predictive value of 18F-DCFPyL PET/CT on a per-region basis, with regions being the prostate or prostate bed, pelvis, extra pelvis, and bones | 3.5 years
  To determine the positive predictive value of 18F-DCFPyL PET/CT on a per-region basis
To determine the sensitivity and specificity of 18F-DCFPyL PET/CT on a per patient and region basis | 3.5 years
  To determine the sensitivity and specificity of 18F-DCFPyL PET/CT on a per patient and region basis

OTHER OUTCOMES:
To characterize ctDNA and exosomes in patients with prostate cancer | 3.5 years
  To characterize ctDNA and exosomes in patients with prostate cancer
To determine correlation with ctDNA and/or exosome levels with disease burden | 3.5 years
  To determine correlation with ctDNA and/or exosome levels with disease burden

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C. Dallos, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No